CLINICAL TRIAL: NCT05969470
Title: Compare the Efficacy of Long-nailed and Short-nailed Fixation for Proximal Femur Metastasis - a Non-inferior Randomized Controlled Trial
Brief Title: Short Versus Long Intramedullary Nails in the Treatment of Proximal Femur Metastasis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other); National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202301173DINA
Record Dates: First submitted 2023-05-09; First posted 2023-08-01 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-05

CONDITIONS: Bone Metastases; Pathological Fracture; Pathological Fracture, Left Femur; Pathological Fracture, Right Femur
Keywords: Long Intramedullary Nails; Short Intramedullary Nails; Bone Metastases; Pathological Fracture of Femur
MeSH Terms: conditions — Fractures, Spontaneous | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Short intramedullary nails (Experimental): The patients receives bone fixation with short intramedullary nails for extremity metastases.
  Interventions: Device: Internal fixation with short intramedullary nails
- Long intramedullary nails (Active Comparator): The patients receives bone fixation with long intramedullary nails for extremity metastases.
  Interventions: Device: Internal fixation with long intramedullary nails

INTERVENTIONS:
Device: Internal fixation with short intramedullary nails — Intramedullary nailing is a method of internal fixation used to treat fractures. An intramedullary nail is a metal rod forced into the marrow canal of a bone to stabilize and align fractures. Participants in this group will be fixed with a shorter intramedullary nail (defined as defined as less than 2/3 of the patient's femur) for proximal femoral (impending) pathological fractures.
  Arms: Short intramedullary nails
Device: Internal fixation with long intramedullary nails — Intramedullary nailing is a method of internal fixation used to treat fractures. An intramedullary nail is a metal rod forced into the marrow canal of a bone to stabilize and align fractures. Participants in this group will be fixed with a longer intramedullary nail (defined as greater than 2/3 of the patient's femur) for proximal femoral (impending) pathological fractures.
  Arms: Long intramedullary nails

SUMMARY:
The goal of this interventional randomized controlled trial is to compare the clinical outcomes in treating extremities pathological fractures (fractures of limbs caused by metastatic tumors) or impending pathological fractures with short or long intramedullary nails. The main questions it aims to answer are:

1. What is the rate of developing new distant metastasis of the operated extremities?
2. Does treating extremities (impending) pathological fractures with long intramedullary nails have lower or similar reoperation rate than the short nails?
3. Are there any differences when comparing the surgical-related complication, functional outcomes and life quality assessment between treating extremities (impending) pathological fractures with long or short intramedullary nails.

Participants who meet surgical indication will be randomized into either the long or short intramedullary nail group after informed consent. The patient will receive bone fixation with the corresponding prosthesis.

DETAILED DESCRIPTION:
Participants will be randomized into either long or short intramedullary nail groups. Participants in the long intramedullary nail group will be fixed with a longer intramedullary nail (defined as greater than 2/3 of the patient's femur) for proximal femoral (impending) pathological fractures, while patients in the short intramedullary nail group will be fixed with a shorter intramedullary nail (defined as less than 2/3 of the patient's femur) for proximal femoral (impending) pathological fractures. Follow-up will be performed at 1, 3, 6, and 12 months after surgery to analyze the patient's function, blood sampling values, and imaging follow-up. The functional capacity will be evaluated by PROMIS questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Femur (impending) pathological fracture that is suitable for intramedullary nail fixation as determined by the physician
* Patient is willing to participate in this clinical trial and cooperate with follow-up

Exclusion Criteria:

* The patient has a more appropriate treatment alternative to single intramedullary nail fixation as determined by the multidisciplinary decision, such as,

  * The metastatic lesions involved the femur head
  * The metastatic lesions involved the pelvis
  * The metastatic lesions compromised the greater or lesser trochanter to a certain extent that arthroplasty was indicated
  * The metastatic lesions involved/occurred more distal than the intertrochanteric line
* There are justified, clinically significant rationales that either long or short intramedullary nails be a more appropriate treatment during pre-operative assessment
* The patient has imaging-confirmed distant femoral metastases before treatment
* Patient has renal cell carcinoma or sarcoma
* Patient is unable to cooperate with follow-up or to understand the trial protocol
* Patient is unable to communicate in Chinese

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-31 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Reoperation rate | Up to 1 year after the intervention
  Percentage of patients receiving revision surgery within 1 year after the intervention. The primary outcome should be compared using non-inferior tests. The non-inferior margin was pre-specified at 25.4%.

SECONDARY OUTCOMES:
Change from baseline in functional outcome on the Patient-Reported Outcomes Measurement Information System-29 scoring at 1,3,6,12 months after the intervention | At 1,3,6,12 months after the intervention
  The Patient-Reported Outcomes Measurement Information System (PROMIS) is a set of person-centered measures that evaluates physical, mental, and social health in adults and children. It's used to measure symptoms and other aspects of health status in a wide variety of chronic diseases. PROMIS-29 is a particular version of this system that covers multiple domains of health and function. It consists of 29 items in total, spanning seven domains: physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, and pain interference. Each domain has four questions, with the exception of the pain interference domain, which has five. Each question is scored from 1-5, the higher score indicates better function or quality of life. The sum of the PROMIS results in the raw score, which lies between 4 and 20. There's also a single question evaluating pain intensity, as assessed by pain intensity numeric rating scale.
Cardiopulmonary complication rate within 30 days after the intervention | Up to 30 days after the intervention
  Cardiopulmonary complication includes the following events developing within 30 days after the intervention: O2 desaturation, shock, embolic event, or coma and death.
Mortality rate at 1,3,6,12 months after the intervention | At 1,3,6,12 months after the intervention
  Percentage of demise at 1,3,6,12 months after the intervention
Percentage of of participants with distant femoral metastasis | Up to 1 year after the intervention
  Newly formed metastatic lesions on the same limb distant to the operation site within 1 year after the intervention
Cost-effectiveness analysis | Up to 2 year after the intervention
  Utility comparison using Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang Chieh Hsieh, MD, Study Chair — Department of Orthopaedic Surgery, National Taiwan University Hospital, Hsin-Chu branch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alvi HM, Damron TA. Prophylactic stabilization for bone metastases, myeloma, or lymphoma: do we need to protect the entire bone? Clin Orthop Relat Res. 2013 Mar;471(3):706-14. doi: 10.1007/s11999-012-2656-1. Epub 2012 Oct 27. PMID 23104043